CLINICAL TRIAL: NCT01816178
Title: Using a Voice Output Communication Aid to Facilitate Language Development in Young Children With Autism Disorders
Brief Title: Using a Voice Output Communication Aid to Facilitate Language Development in Young Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, Dennis Campbell, Associate Professor, University of South Alabama
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASUIRB-1
Record Dates: First submitted 2013-03-11; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Autistic Disorder
Keywords: Autism spectrum Disorders; Voice Output Communication
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- communication training (Experimental): Participants were instructed in the use of a voices output communication aid.
  Interventions: Behavioral: communication training

INTERVENTIONS:
Behavioral: communication training — Participants were instructed in the use of a voices output communication aid.

SUMMARY:
It was proposed that in order to teach these children to use a Voice Output Communication Aid (VOCA), it should be introduced through a play-based situation using parents as the primary interventionist.

DETAILED DESCRIPTION:
The research will test the effectiveness of using the communication board to improve the frequency of communication and social engagement for these children, and the level or sophistication of that engagement. The study will test the effectiveness of using the communication board in a variety of settings and a variety of practitioners. The study will have sites in and near Jonesboro, Arkansas.

ELIGIBILITY:
Inclusion Criteria:

Criteria for inclusion included a diagnosis of autism and agreement of the parents to participate and use the VOCA at home.

Exclusion Criteria:

Not diagnosed with Autism Spectrum disorder

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2004-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Improved Communication | 1 year
  Surveys of number of words Text data from VOCA Formal assessment instruments

SECONDARY OUTCOMES:
Review of text output from the VOCA | 1 year
  The VOCA records data on usage by day and time. We analyze the text data from the VOCA.

OTHER OUTCOMES:
Improved parent interaction | 1 year
  Data were gathered from the parents on the number of words spoken by their son and the way they "felt" the intervention was proceeding. Essentially we had parents report on the effectiveness of using the VOCA to improve the frequency of communication and social engagement for these young children with ASD.

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas State University, State University, Arkansas, United States